CLINICAL TRIAL: NCT01613118
Title: Efficacy and Safety of Sparsentan (RE-021), a Dual Endothelin Receptor and Angiotensin Receptor Blocker, in Patients With Focal Segmental Glomerulosclerosis (FSGS): a Randomized, Double-Blind, Active-Control, Dose-Escalation Study
Brief Title: Randomized, Double-Blind, Safety and Efficacy Study of RE-021 (Sparsentan) in Focal Segmental Glomerulosclerosis
Acronym: DUET
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Travere Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RET-D-001; NCT01622738 (obsolete NCT alias)
Record Dates: First submitted 2012-06-04; First posted 2012-06-06 (Estimated); Results first posted 2021-07-27 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-04

CONDITIONS: Focal Segmental Glomerulosclerosis
Keywords: Primary FSGS; Nephrotic syndrome; Steroid Resistant
MeSH Terms: conditions — Glomerulosclerosis, Focal Segmental; Nephrotic Syndrome | interventions — sparsentan; Irbesartan

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- RE-021 (Sparsentan) 200 mg - Double-Blind Period (Experimental): RE-021 (Sparsentan) will be administered as a single oral morning dose. In this ARM the RE-021 (Sparsentan) dose will be 200mg.
  Patients at </= 50kg will receive half of the RE-021 (Sparsentan) dose for the 8 week duration.
  Interventions: Drug: RE-021 (Sparsentan)
- RE-021 (Sparsentan) 400 mg - Double-Blind Period (Experimental): RE-021 (Sparsentan) will be administered as a single oral morning dose. In this ARM the RE-021 (Sparsentan) dose will be 400mg.
  Patients at </= 50kg will receive half of the RE-021 (Sparsentan) dose for the 8 week duration.
  Interventions: Drug: RE-021 (Sparsentan)
- RE-021 (Sparsentan) 800 mg - Double-Blind Period (Experimental): RE-021 (Sparsentan) will be administered as a single oral morning dose. In this ARM the RE-021 (Sparsentan) dose will be 800mg.
  Patients at </= 50kg will receive half of the RE-021 (Sparsentan) dose for the 8 week duration.
  Interventions: Drug: RE-021 (Sparsentan)
- Irbesartan 300 mg - Double-Blind Period (Active Comparator): The control will be administered irbesartan as a single oral dose of 150mg for the first week before escalating to 300mg for the remaining 7 weeks.
  Patients at </= 50kg will receive 150mg irbesartan for the 8 week duration.
  Interventions: Drug: Irbesartan
- RE-021 (Sparsentan) - Open-Label Extension Period (Experimental): Includes all subjects who completed the Double-Blind period and enrolled in the Open-Label Extension period of the study.
  All subjects who completed the Double-Blind period were evaluated for response and safety at the Week 8 visit to determine eligibility for continued treatment on their assigned doses in an Open-Label Extension period for up to 496 additional weeks. Subjects treated with irbesartan during the Double-Blind period were offered sparsentan treatment at the dose they would have received according to the Double-Blind dose cohort in which they were enrolled.
  Interventions: Drug: RE-021 (Sparsentan)

INTERVENTIONS:
Drug: RE-021 (Sparsentan) — Oral, once-daily
  Other Names: Sparsentan
  Arms: RE-021 (Sparsentan) - Open-Label Extension Period; RE-021 (Sparsentan) 200 mg - Double-Blind Period; RE-021 (Sparsentan) 400 mg - Double-Blind Period; RE-021 (Sparsentan) 800 mg - Double-Blind Period
Drug: Irbesartan — Oral, once-daily
  Other Names: Avapro
  Arms: Irbesartan 300 mg - Double-Blind Period

SUMMARY:
This study will investigate whether RE-021 (Sparsentan), a selective dual-acting receptor antagonist with affinity for endothelin (A type) and angiotensin II receptors (Type 1), is safe and effective in treating patients with focal segmental glomerulosclerosis (FSGS).

DETAILED DESCRIPTION:
Focal segmental glomerulosclerosis (FSGS) is a rare glomerular disorder which results in frank proteinuria and in some patients progression to end-stage kidney disease (ESKD) over 5-10 years. Proteinuria reduction is widely regarded to be beneficial and is considered the primary goal of treatment in FSGS and slowing its progressive course (D'Agati, et. al, 2011). Patients are currently treated with angiotensin receptor blockers (ARB) and angiotensin converting inhibitors (ACEI) to lower proteinuria with steroids, calcineurin inhibitors, and other immunosuppressive agents reserved for patients with severe proteinuria and in particular with nephrotic syndrome. Despite these therapies, many patients have nephrotic range proteinuria and new therapeutic agents are needed. Endothelin receptor antagonists (ERA) have been shown to lower proteinuria in clinical trials of diabetic nephropathy and have been speculated to be effective in FSGS.

ELIGIBILITY:
Inclusion Criteria

1. Biopsy-proven FSGS OR documentation of a genetic mutation in a podocyte protein associated with the disease.
2. Urine protein/creatinine ratio (Up/C) at or above 1.0 g/g.
3. Estimated glomerular filtration rate (eGFR) >30.
4. Mean seated blood pressure (BP) >100/60 mmHg and <145/95 in patients >/= 18 years of age. Mean seated BP for patients <18 years of age should be >90/60 mmHg and <95th percentile for age, gender, and height.
5. If a patient is taking immunosuppressive medications (except for Rituximab or cyclophosphamide), the dose and/or levels must be stable for 1 month prior to randomization and the Investigator should not have plans to alter the regimen during the first 8 weeks of treatment, except to stabilize levels. Patients on Rituximab or cyclophosphamide will be eligible provided they have not been taking these medications for 3 months prior to randomization.
6. US Sites: Males or females 8 to 75 years of age willing and able to provide written informed consent and/or assent, with informed consent signed by patient or parent/legal guardian.
7. EU Sites: Males or females 18 to 75 years of age willing and able to provide written informed consent, with informed consent, signed by patient or legal guardian.

Exclusion Criteria

1. Patients with FSGS secondary to another condition.
2. Patients with history of type 1 diabetes mellitus, uncontrolled type 2 diabetes mellitus (HBA1c>8%), or non-fasting blood glucose >180 mg/dL at screening.
3. Patients who have had any organ transplant.
4. Patients with a requirement for any of the medications indicated on the list of Excluded Medications, with the exception of ACE and ARBs.
5. Patients with a documented history of heart failure (NYHA Class II-IV), and / or previous hospitalization for heart failure or unexplained dyspnea, orthopnea, paroxysmal nocturnal dyspnea, ascites and peripheral edema. Patients with clinically significant cerebrovascular disease (transient ischemic attack or stroke) and/or coronary artery disease (hospitalization for myocardial infarction or unstable angina, new onset of angina with positive functional tests or coronary angiogram revealing stenosis, coronary revascularization procedure) within 6 months before screening.
6. Patients with clinically significant cardiac conduction defects, including second or third degree atrioventricular block, left bundle branch block, sick sinus syndrome, atrial fibrillation, atrial flutter, an accessory bypass tract, or any arrhythmia requiring medication.
7. Patients with jaundice, hepatitis, or known hepatobiliary disease (includes asymptomatic cholelithiasis); alanine aminotransferase and/or aspartate aminotransferase >2 times the upper limit of normal at Screening.
8. Patients positive for human immunodeficiency virus (HIV), and markers indicating acute (positivity of at least one of the following: Hepatitis B surface antigen [HBsAg], Hepatitis B "e" antigen [HBeAg], Hepatitis B virus [HBV] DNA in blood or liver, Immunoglobulin M Hepatitis B core antibody) or chronic (HBsAg and/or HBeAg and/or Hepatitis B virus [HBV] DNA positivity) HBV infection, or hepatitis C virus (HCV) infection (reactive anti-HCV antibody and/or HCV RNA). Testing at screening is only required for patients >/= 18 years of age.
9. History of malignancy other than adequately treated basal cell or squamous cell skin cancer within the past 5 years.
10. Patients with hemodynamically significant valvular disease.
11. Hematocrit (HCT) <27 or hemoglobin (Hgb) <9.
12. Potassium >5.5 mEq/L.
13. Patients >18 years of age with Estimated Glomerular Filtration Rate (eGFR) ≥60 ml mL/min who have N-terminal prohormone of brain natriuretic peptide (NT-proBNP) ≥200 pg/mL (57.8 pmol/L). For patients >18 years of age with eGFR <60 mL/min, the following parameters requiring echocardiography (ECHO) at screening should be used for exclusion:

    1. NT-proBNP ≥300 pg/mL in patients >18 years of age with eGFR 45 59.9 mL/min
    2. NT-proBNP = 200-299 pg/mL in patients >18 years of age with eGFR 45 59.9 mL/min, and abnormal ejection fraction (EF <55) and/or diastolic dysfunction on ECHO
    3. NT-proBNP ≥400 pg/mL in patients >18 years of age with eGFR 30.0 44.9 mL/min
    4. NT-proBNP = 200-399 pg/mL in patients >18 years of age with eGFR 30.0 44.9 mL/min, and abnormal ejection fraction (EF <55) and/or diastolic dysfunction on ECHO.
14. Patients >/= 18 years of age with body mass index (BMI) >40. Patients <18 years of age with a BMI in the 99% percentile plus 5 units.
15. Patients who have abnormal clinical laboratory values at Screening, which are designated by the Principal Investigator as clinically significant.
16. Patients with a history of drug or alcohol abuse within the past two years.
17. Patients with a history of an allergic response to any angiotensin II antagonist or endothelin receptor antagonist.
18. Women who are pregnant or breastfeeding.
19. Women of child-bearing potential (WOCBP) who are unwilling or unable to use two reliable methods of contraception, with at least one being highly reliable (e.g. oral, implanted or injected contraceptive hormones or an intrauterine device) and one being a barrier method, in order to avoid pregnancy for the entire study period and for 90 days post study participation. WOCBP, defined as all women physiologically capable of becoming pregnant, includes any female who has experienced menarche and who has not undergone successful surgical sterilization (hysterectomy, bilateral tubal ligation or bilateral ovariectomy) or is not postmenopausal (defined as amenorrhea >12 consecutive months and for women on hormone replacement therapy, only with documented plasma follicle stimulating hormone level greater than 35 mIU/mL). Women using oral, implanted or injected contraceptive hormones, an intrauterine device, barrier methods (diaphragm, condoms, spermicidal) to prevent pregnancy, practicing abstinence or where the partner is sterile (e.g. vasectomy) As well as postmenopausal women who have fertilized eggs implanted are also considered WOCBP.
20. Patients who have participated in another investigational drug study within 28 days prior to screening, or who will participate in another drug study during the course of this study.
21. Prior exposure to Sparsentan, dual acting receptor antagonist (DARA), or PS433540.
22. Patients who are unable to comply with the study procedures and assessments, including the ability swallow the study drug or control capsules.

Ages: 8 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2014-03 (Actual); Primary Completion 2016-06 (Actual); Study Completion 2024-03-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Howard Trachtman, M.D., Principal Investigator — NYU School of Medicine
Locations (33):
- United States (28):
  - Balboa Nephrology Medical Group, San Diego, California
  - Los Angeles Biomedical Research Institute, Torrance, California
  - Colorado Kidney Care, Denver, Colorado
  - University of Miami Miller School of Medicine, Miami, Florida
  - Miami Children's Hospital, Miami, Florida
  - University of Iowa Children's Hospital, Iowa City, Iowa
  - Renal and Transplant Associates of New England, PC, Springfield, Massachusetts
  - University of Minnesota, Minneapolis, Minnesota
  - The Children's Mercy Hospital, Kansas City, Missouri
  - NYU Langone Medical Center, New York, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Columbia University Medical Center, New York, New York
  - SUNY Stony Brook Hospital, Stony Brook, New York
  - UNC Kidney Center, Pediatrics, Chapel Hill, North Carolina
  - University North Carolina (UNC) Kidney Center, Chapel Hill, North Carolina
  - Akron Nephrology Associates, Akron, Ohio
  - The Cleveland Clinic Foundation, Cleveland, Ohio
  - Unversity of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Northeast Clinical Research Center, Bethlehem, Pennsylvania
  - The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Temple University School of Medicine, Philadelphia, Pennsylvania
  - University of Pennsylvania, Perelman School of Medicine, Philadelphia, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Clinical Advancement Center, San Antonio, Texas
  - Southern Utah Kidney and Hypertension Center, St. George, Utah
  - University of Washington, Seattle, Washington
  - Catholic Health Initiatives Franciscan, Tacoma, Washington
  - Marshfield Clinic Research Foundation, Marshfield, Wisconsin
- General Teaching Hospital Prague, Prague, Czechia
- Italy (4):
  - Azienda Ospedaliero Universitaria Policlinico di Bari, Bari
  - Azienda Ospedaliero Universitaria Careggi, Florence
  - IRCCS Istituti Clinici Maugeri, Pavia
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Rome

REFERENCES:
- [Background] D'Agati VD, Kaskel FJ, Falk RJ. Focal segmental glomerulosclerosis. N Engl J Med. 2011 Dec 22;365(25):2398-411. doi: 10.1056/NEJMra1106556. No abstract available. PMID 22187987
- [Result] Campbell KN, Gesualdo L, Murphy E, Rheault MN, Srivastava T, Tesar V, Komers R, Trachtman H. Sparsentan for Focal Segmental Glomerulosclerosis in the DUET Open-Label Extension: Long-term Efficacy and Safety. Kidney Med. 2024 Apr 26;6(6):100833. doi: 10.1016/j.xkme.2024.100833. eCollection 2024 Jun. PMID 38831932
- [Result] Trachtman H, Nelson P, Adler S, Campbell KN, Chaudhuri A, Derebail VK, Gambaro G, Gesualdo L, Gipson DS, Hogan J, Lieberman K, Marder B, Meyers KE, Mustafa E, Radhakrishnan J, Srivastava T, Stepanians M, Tesar V, Zhdanova O, Komers R; DUET Study Group. DUET: A Phase 2 Study Evaluating the Efficacy and Safety of Sparsentan in Patients with FSGS. J Am Soc Nephrol. 2018 Nov;29(11):2745-2754. doi: 10.1681/ASN.2018010091. PMID 30361325
- [Derived] Liu ID, Willis NS, Craig JC, Hodson EM. Interventions for idiopathic steroid-resistant nephrotic syndrome in children. Cochrane Database Syst Rev. 2025 May 8;5(5):CD003594. doi: 10.1002/14651858.CD003594.pub7. PMID 40337980
- [Derived] Omachi K, O'Carroll C, Miner JH. PPAR delta Agonism Ameliorates Renal Fibrosis in an Alport Syndrome Mouse Model. Kidney360. 2023 Mar 1;4(3):341-348. doi: 10.34067/KID.0006662022. PMID 36657027
- [Derived] Hodson EM, Sinha A, Cooper TE. Interventions for focal segmental glomerulosclerosis in adults. Cochrane Database Syst Rev. 2022 Feb 28;2(2):CD003233. doi: 10.1002/14651858.CD003233.pub3. PMID 35224732

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: For the Double-Blind (DB) period, patients were screened to confirm eligibility and underwent 2-wk washout period to discontinue ARBs or ACEIs if necessary. Subjects who completed DB period were evaluated to determine eligibility for the Open-Label Extension (OLE) period (up to 496 additional weeks), those treated with irbesartan were offered sparsentan in the OLE period. Dose changes were permitted during the OLE so all subjects enrolled in OLE are included in RE-021(Sparsentan)-OLE Period arm.
Groups:
- RE-021 (Sparsentan) 200 mg - Double-Blind Period: RE-021 (Sparsentan) administered as a single oral morning dose. In this ARM the RE-021 (Sparsentan) dose was 200mg.
  Patients at </= 50kg received half the RE-021 (Sparsentan) dose for the 8 week duration.
  RE-021 (Sparsentan): Oral, once-daily
- RE-021 (Sparsentan) 400 mg - Double-Blind Period: RE-021 (Sparsentan) administered as a single oral morning dose. In this ARM the RE-021 (Sparsentan) dose was 400mg.
  Patients at </= 50kg received half the RE-021 (Sparsentan) dose for the 8 week duration.
  RE-021 (Sparsentan): Oral, once-daily
- RE-021 (Sparsentan) 800 mg - Double-Blind Period: RE-021 (Sparsentan) administered as a single oral morning dose. In this ARM the RE-021 (Sparsentan) dose was 800mg.
  Patients at </= 50kg received half of the RE-021 (Sparsentan) dose for the 8 week duration.
  RE-021 (Sparsentan): Oral, once-daily
- Irbesartan 300 mg - Double-Blind Period: The control irbesartan was administered as a single oral dose of 150mg for the first week before being escalated to 300mg for the remaining 7 weeks.
  Patients at </= 50kg received 150mg irbesartan for the 8 week duration.
  Irbesartan: Oral, once-daily
- RE-021 (Sparsentan) - Open-Label Extension Period: Includes all subjects who completed the Double-Blind period and enrolled in the Open-Label Extension period of the study.
  All subjects who completed the Double-Blind period were evaluated for response and safety at the Week 8 visit to determine eligibility for continued treatment on their assigned doses in an Open-Label Extension period for up to 496 additional weeks. Subjects treated with irbesartan during the Double-Blind period were offered sparsentan treatment at the dose they would have received according to the Double-Blind dose group in which they were enrolled.
  Sparsentan (RE-021): Oral, once-daily
Period: Double-blind
Arm/Group | RE-021 (Sparsentan) 200 mg - Double-Blind Period | RE-021 (Sparsentan) 400 mg - Double-Blind Period | RE-021 (Sparsentan) 800 mg - Double-Blind Period | Irbesartan 300 mg - Double-Blind Period | RE-021 (Sparsentan) - Open-Label Extension Period
Started | 13 | 26 | 34 | 36 | 0 (Subjects are shown in the respective double-blind arm.)
Completed | 13 | 23 | 32 | 35 | 0 (Subjects are shown in the respective double-blind arm.)
Not Completed | 0 | 3 | 2 | 1 | 0
Period: Open-label Extension
Arm/Group | RE-021 (Sparsentan) 200 mg - Double-Blind Period | RE-021 (Sparsentan) 400 mg - Double-Blind Period | RE-021 (Sparsentan) 800 mg - Double-Blind Period | Irbesartan 300 mg - Double-Blind Period | RE-021 (Sparsentan) - Open-Label Extension Period
Started | 0 (All subjects who completed the Double-Blind period and enrolled in the Open-Label Extension period of the study are captured in the "RE-021 (Sparsentan) - Open-Label Extension Period" arm.) | 0 (All subjects who completed the Double-Blind period and enrolled in the Open-Label Extension period of the study are captured in the "RE-021 (Sparsentan) - Open-Label Extension Period" arm.) | 0 (All subjects who completed the Double-Blind period and enrolled in the Open-Label Extension period of the study are captured in the "RE-021 (Sparsentan) - Open-Label Extension Period" arm.) | 0 (All subjects who completed the Double-Blind period and enrolled in the Open-Label Extension period of the study are captured in the "RE-021 (Sparsentan) - Open-Label Extension Period" arm.) | 103 (All subjects who completed the Double-Blind period and enrolled in the Open-Label Extension period of the study are captured in the "RE-021 (Sparsentan) - Open-Label Extension Period" arm.)
Active at Study End (At the time the study ended, thirty subjects were participating in the study but had not yet completed 496 weeks in the open-label extension period.) | 0 | 0 | 0 | 0 | 30
Completed | 0 | 0 | 0 | 0 | 1
Not Completed | 0 | 0 | 0 | 0 | 102

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | RE-021 (Sparsentan) 200 mg - Double-Blind Period | RE-021 (Sparsentan) 400 mg - Double-Blind Period | RE-021 (Sparsentan) 800 mg - Double-Blind Period | Irbesartan 300 mg - Double-Blind Period | Total
Number analyzed (Participants) | 13 | 26 | 34 | 36 | 109
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.8 (14.36) | 38.3 (16.78) | 35.9 (17.68) | 34.1 (15.96) | 36.7 (16.54)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 9 | 17 | 17 | 49
  Male | 7 | 17 | 17 | 19 | 60

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in Urine Protein/Creatinine (Up/C)
Description: Primary efficacy objective is to determine the change in UP/C in FSGS patients receiving RE-021 (Sparsentan) from baseline to 8 weeks over a range of dose levels compared to treatment with irbesartan as active control.
Time Frame: 8 weeks
Population: Efficacy evaluable set
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: percent change
Groups:
- RE-021 (Sparsentan) 200, 400, 800 mg Pooled: RE-021 (Sparsentan) administered as a single oral morning dose. In this ARM the RE-021 (Sparsentan) dose was 200, 400, or 800mg.
  Patients at </= 50kg received half of the RE-021 (Sparsentan) dose for the 8 week duration.
  RE-021 (Sparsentan): Oral, once-daily
- Irbesartan 300 mg Pooled: The control irbesartan was administered as a single oral dose of 150mg for the first week before being escalated to 300mg for the remaining 7 weeks.
  Patients at </= 50kg received 150mg irbesartan for the 8 week duration.
  Irbesartan: Oral, once-daily
- RE-021 (Sparsentan) 400 and 800 mg Pooled: RE-021 (Sparsentan) administered as a single oral morning dose. In this ARM the RE-021 (Sparsentan) dose was 400 or 800mg.
  Patients at </= 50kg received half of the RE-021 (Sparsentan) dose for the 8 week duration.
  RE-021 (Sparsentan): Oral, once-daily
- RE-021 (Sparsentan) 200mg: RE-021 (Sparsentan) administered as a single oral morning dose. In this group, the RE-021 (Sparsentan) dose was 200mg.
  Patients at </= 50kg received half of the RE-021 (Sparsentan) dose for the 8 week duration.
  RE-021 (Sparsentan): Oral, once-daily
- RE-021 (Sparsentan) 400mg: RE-021 (Sparsentan) administered as a single oral morning dose. In this group, the RE-021 (Sparsentan) dose was 400mg.
  Patients at </= 50kg received half of the RE-021 (Sparsentan) dose for the 8 week duration.
  RE-021 (Sparsentan): Oral, once-daily
- RE-021 (Sparsentan) 800mg: RE-021 (Sparsentan) administered as a single oral morning dose. In this group, the RE-021 (Sparsentan) dose was 800mg.
  Patients at </= 50kg received half of the RE-021 (Sparsentan) dose for the 8 week duration.
  RE-021 (Sparsentan): Oral, once-daily
Arm/Group | RE-021 (Sparsentan) 200, 400, 800 mg Pooled | Irbesartan 300 mg Pooled | RE-021 (Sparsentan) 400 and 800 mg Pooled | RE-021 (Sparsentan) 200mg | RE-021 (Sparsentan) 400mg | RE-021 (Sparsentan) 800mg
Number analyzed (Participants) | 64 | 32 | 51 | 13 | 21 | 30
percent change | -44.8 [-52.7 to -35.7] | -18.5 [-34.6 to 1.7] | -47.4 [-56.3 to -36.9] | -33.1 [-49.3 to -11.6] | -52.7 [-64.3 to -37.2] | -41.3 [-54.4 to -24.4]

2. Secondary Outcome: Percentage of Patients Achieving FSGS Partial Remission Endpoint (FPRE)
Description: The secondary efficacy endpoint is the proportion of FSGS patients achieving FPRE (experiencing a UP/C ratio ≤1.5 g/g and >40% reduction from baseline in Up/C) at Week 8 over a range of dose levels compared to treatment with irbesartan as active control.
Time Frame: 8 weeks
Population: Efficacy evaluable set. The sparsentan arms were compared to irbesartan in several different combinations that were defined in the study's Statistical Analysis Plan.
Measure: Number; unit: percentage of patients
Groups:
- RE-021 (Sparsentan) 200 mg: RE-021 (Sparsentan) administered as a single oral morning dose. In this group, the RE-021 (Sparsentan) dose was 200mg.
  Patients at </= 50kg received half of the RE-021 (Sparsentan) dose for the 8 week duration.
  RE-021 (Sparsentan): Oral, once-daily
- RE-021 (Sparsentan) 400 mg: RE-021 (Sparsentan) administered as a single oral morning dose. In this group, the RE-021 (Sparsentan) dose was 400mg.
  Patients at </= 50kg received half of the RE-021 (Sparsentan) dose for the 8 week duration.
  RE-021 (Sparsentan): Oral, once-daily
- RE-021 (Sparsentan) 800 mg: RE-021 (Sparsentan) administered as a single oral morning dose. In this group, the RE-021 (Sparsentan) dose was 800mg.
  Patients at </= 50kg received half of the RE-021 (Sparsentan) dose for the 8 week duration.
  RE-021 (Sparsentan): Oral, once-daily
Arm/Group | RE-021 (Sparsentan) 200, 400, 800 mg Pooled | Irbesartan 300 mg Pooled | RE-021 (Sparsentan) 400 and 800 mg Pooled | RE-021 (Sparsentan) 200 mg | RE-021 (Sparsentan) 400 mg | RE-021 (Sparsentan) 800 mg
Number analyzed (Participants) | 64 | 32 | 51 | 13 | 21 | 30
percentage of patients | 28.13 | 9.38 | 31.37 | 15.38 | 38.10 | 26.67

ADVERSE EVENTS:
Time Frame: For double-blind treatment arms: 8 weeks. For all sparsentan analysis including the open-label extension period: up to 508 weeks.
Description: Adverse Events are reported for each treatment arm in the Double-Blind period and for sparsentan-treated patients across the entire study (Double-Blind and Open-Label Extension periods). As one objective of the study was to evaluate the long-term safety of sparsentan, the sparsentan safety results for the entire study are presented in the "All Sparsentan (Double-Blind and Open-Label Extension)" reporting group as pre-specified in the study's Statistical Analysis Plan.
Groups:
- RE-021 (Sparsentan) 200 mg - Double-Blind Period: Sparsentan (RE-021) administered as a single oral morning dose. In this ARM the sparsentan (RE-021) dose was 200mg.
  Patients at </= 50kg received half the sparsentan (RE-021) dose for the 8 week duration.
  Sparsentan (RE-021): Oral, once-daily
- RE-021 (Sparsentan) 400 mg - Double-Blind Period: Sparsentan (RE-021) administered as a single oral morning dose. In this ARM the sparsentan (RE-021) dose was 400mg.
  Patients at </= 50kg received half the sparsentan (RE-021) dose for the 8 week duration.
  Sparsentan (RE-021): Oral, once-daily
- RE-021 (Sparsentan) 800 mg - Double-Blind Period: Sparsentan (RE-021) administered as a single oral morning dose. In this ARM the sparsentan (RE-021) dose was 800mg.
  Patients at </= 50kg received half of the sparsentan (RE-021) dose for the 8 week duration.
  Sparsentan (RE-021): Oral, once-daily
- Irbesartan 300 mg - Double-Blind Period: The control irbesartan was administered as a single oral dose of 150mg for the first week before escalating to 300mg for the remaining 7 weeks.
  Patients at </= 50kg received 150mg irbesartan for the 8 week duration.
  Irbesartan: Oral, once-daily
- All Sparsentan (Double-Blind and Open-Label Extension): Double-blind and open-label extension data for all patients while on sparsentan (RE-021). This includes double-blind and open-label extension data for subjects randomized to sparsentan, and only open-label extension data for subjects randomized to irbesartan.
  Sparsentan (RE-021): Oral, once-daily
Arm/Group | RE-021 (Sparsentan) 200 mg - Double-Blind Period | RE-021 (Sparsentan) 400 mg - Double-Blind Period | RE-021 (Sparsentan) 800 mg - Double-Blind Period | Irbesartan 300 mg - Double-Blind Period | All Sparsentan (Double-Blind and Open-Label Extension)
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/26 | 0/34 | 0/36 | 0/108
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/26 | 2/34 | 1/36 | 48/108
Other Adverse Events (participants affected / at risk) | 11/13 | 17/26 | 27/34 | 26/36 | 104/108
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RE-021 (Sparsentan) 200 mg - Double-Blind Period (N=13) | RE-021 (Sparsentan) 400 mg - Double-Blind Period (N=26) | RE-021 (Sparsentan) 800 mg - Double-Blind Period (N=34) | Irbesartan 300 mg - Double-Blind Period (N=36) | All Sparsentan (Double-Blind and Open-Label Extension) (N=108)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 10 (11)
Proteinuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
End stage renal disease (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Chronic kidney disease (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nephrotic syndrome (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Renal impairment (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Subcapsular renal haematoma (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 10 (11)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Abscess limb (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Septic shock (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Chest discomfort (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Drug withdrawal syndrome (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Generalised oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypervolaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anal fistula (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Erosive oesophagitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Melaena (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Angiopathy (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haematoma (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypertensive urgency (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Jugular vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Aortic valve stenosis (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Conduction disorder (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Coronary artery stenosis (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Supraventricular extrasystoles (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bone infarction (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Alcohol poisoning (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Jaw fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Angioimmunoblastic T-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3)
Apnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Glomerular filtration rate decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pulse absent (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Endometrial hyperplasia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ovarian cyst (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperaldosteronism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Liver injury (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RE-021 (Sparsentan) 200 mg - Double-Blind Period (N=13) | RE-021 (Sparsentan) 400 mg - Double-Blind Period (N=26) | RE-021 (Sparsentan) 800 mg - Double-Blind Period (N=34) | Irbesartan 300 mg - Double-Blind Period (N=36) | All Sparsentan (Double-Blind and Open-Label Extension) (N=108)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 17 (19)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (3) | 2 (2) | 17 (43)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 13 (23)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 11 (22)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 9 (10)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 8 (11)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 7 (10)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 6 (6)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 6 (6)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 4 (4) | 1 (1) | 27 (36)
Nausea (Gastrointestinal disorders) | 1 (1) | 3 (3) | 5 (6) | 3 (3) | 26 (37)
Vomiting (Gastrointestinal disorders) | 0 (0) | 3 (3) | 3 (5) | 1 (1) | 19 (30)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 7 (10)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1) | 3 (3) | 2 (2) | 6 (7)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 6 (6)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 5 (6)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Oedema peripheral (General disorders) | 1 (1) | 2 (2) | 2 (2) | 1 (1) | 30 (45)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 16 (19)
Fatigue (General disorders) | 0 (0) | 1 (1) | 2 (3) | 4 (4) | 12 (15)
Chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 10 (14)
Asthenia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 6 (8)
Oedema (General disorders) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 4 (4)
Local swelling (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 17 (21)
Blood creatinine increased (Investigations) | 1 (2) | 1 (1) | 1 (1) | 1 (1) | 16 (23)
Glomerular filtration rate decreased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 11 (15)
Haemoglobin decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 7 (7)
N-terminal prohormone brain natriuretic peptide increased (Investigations) | 0 (0) | 1 (3) | 1 (1) | 0 (0) | 6 (8)
Blood triglycerides increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 3 (5)
Blood potassium increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Headache (Nervous system disorders) | 3 (4) | 2 (2) | 9 (11) | 7 (7) | 32 (43)
Dizziness (Nervous system disorders) | 0 (0) | 4 (4) | 6 (6) | 4 (4) | 19 (28)
Paraesthesia (Nervous system disorders) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 5 (5)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 19 (28)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 14 (15)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 11 (13)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 10 (15)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 7 (8)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 6 (7)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 6 (6)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (3) | 22 (41)
Gout (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 15 (29)
Metabolic acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 10 (12)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 6 (7)
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 6 (6)
Hypotension (Vascular disorders) | 1 (1) | 3 (3) | 6 (6) | 3 (3) | 23 (38)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 19 (30)
Orthostatic hypotension (Vascular disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 4 (5)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 15 (22)
Proteinuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 15 (21)
Renal impairment (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 6 (7)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 7 (8)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 6 (9)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 2 (2) | 2 (3) | 13 (18)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 4 (4) | 12 (17)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 11 (18)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 8 (8)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 7 (9)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 6 (6)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Rash papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 19 (20)
Oligomenorrhoea (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 11 (11)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 3 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes